CLINICAL TRIAL: NCT00977093
Title: A Multicenter, Phase III, Open-label Study of Gadodiamide Injection in Myocardial Perfusion Magnetic Resonance Imaging
Brief Title: A Study of Gadodiamide Injection in Myocardial Perfusion Magnetic Resonance Imaging
Acronym: MR-IMPACT-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amersham Buchler, GmbH & Co KG (Industry)
Collaborators: Beacon Bioscience, Inc. (Industry); The Cleveland Clinic (Other); CRL, Medinet Europe, Breda, The Netherlands (Corelab for blood sample analyses) (Unknown); Biomedical Systems (Industry)
Responsible Party: Prof. Juerg Schwitter, University Hospital Lausanne - CHUV, Switzerland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SOV 303 / SOV 304
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Cardiac magnetic resonance imaging; single photon emission computed tomography; invasive coronary angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perfusion CMR examination (Experimental): All patients will undergo perfusion CMR examination, single-photon emission computed tomography, and conventional invasive coronary angiography.
  Interventions: Other: Perfusion CMR for detection of coronary artery disease; Other: Perfusion cardiac magnetic resonance imaging

INTERVENTIONS:
Other: Perfusion CMR for detection of coronary artery disease — Perfusion CMR is performed during adenosine infusion for vasodilation (3 minutes of 0.14mg/kg/min IV) and injection of Gd-DTPA-BMA at 0.075mmol/kg IV.
  Other Names: MR contrast medium: Gd-DTPA-BMA is Omniscan
Other: Perfusion cardiac magnetic resonance imaging — Perfusion CMR with Gd-DTPA-BMA to detect coronary artery disease
  Other Names: Conventional MR contast medium: Gd-DTPA-BMA is Omniscan

SUMMARY:
The purpose of this study is to determine how well perfusion cardiac magnetic resonance (MR) imaging is able to detect certain heart abnormalities, such as a coronary artery narrowing.

To this purpose, a conventional MR contrast medium (Gd-DTPA-BMA) will be used during an adenosine infusion (an approved substance which enlarges the arteries of the heart, so that the blood flow to the heart muscle increases). This magnetic resonance imaging technique will be compared with single photon emission computed tomography (SPECT), a well-established technique to detect this heart abnormalities.

Both, cardiac MR and SPECT will be compared with invasive coronary angiography, a technique which directly visualized the heart vessels and narrowings of these (=standard of reference).

DETAILED DESCRIPTION:
This study is a multicentre, open label, phase III study in adult subjects designed to show that Gd-DTPA-BMA (a conventional MR contrast medium = OMNISCAN) enhanced myocardial MR perfusion imaging is non-inferior to myocardial SPECT. Both imaging techniques will be performed during adenosine stress (0.14mg/min/kg over 3 minutes IV). Gd-DTPA-BMA will be used twice (2 doses of 0.075 mmol/kg for the stress and rest study each) for the detection of myocardial perfusion defects. The standard of reference is invasive coronary angiography, which defines the presence of coronary artery disease, if vessels of at least 2mm in diameter show stenosis of at least 50% (diameter reduction). Patients with a history of myocardial infarction(s) are positive for coronary artery disease, even when coronary arteries are not stenosed as evidenced by the coronary angiography performed in the setting of this trial(= assigning patients as positive for coronary artery disease after successful PCI-revascularization of acute infarct(s) in the past).

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a man or woman and is 18 years of age or older.
2. For women of childbearing potential, the results of a urine or serum human chorionic gonadotropin (beta-HCG) pregnancy test, done at screening (with the result known before investigational product administration), must be negative. Only those women who are surgically sterile (have had a documented bilateral oophorectomy and/or documented hysterectomy) or postmenopausal (cessation of menses for more than 1 year) will be allowed to enrol in the study without a pregnancy test at screening.
3. The subject is conscious and able to comply with study procedures.
4. Written, informed consent is obtained.
5. The subject is suspected, as a results of their clinical signs and symptoms, of having CAD (most subjects will probably be included using these criteria).
6. The subject is referred to a quantitative CXA for known or suspected CAD or has undergone quantitative CXA within 4 weeks prior to MRI without any intervention or change of symptoms since the CXA examination.
7. The subject is referred for a SPECT for a functional evaluation of myocardial perfusion or has undergone SPECT within 4 weeks prior to MRI without any intervention, or change in symptoms, between the 2 examinations (the findings of SPECT will not be taken into account for inclusion purposes).

Exclusion Criteria:

1. The subject is lactating.
2. The subject is pregnant as defined by a urine or serum beta-HCG pregnancy test obtained within the 24 hours before dosing.
3. The subject was previously included in this study.
4. The subject received an investigational product in the 30 days before or will receive one during or in the 30 days after investigational product administration.
5. The subject has known allergies or a contra-indication to the investigational product.
6. The subject presents any clinically active, serious, life-threatening disease, with a life expectancy of less than 1 month.
7. The subject received or is scheduled to receive an MRI contrast medium (other than the investigational product) within 24 hours prior to or in the 24 hours following the investigational product administration.
8. The subject received or is scheduled to receive an X-ray contrast medium within 12 hours prior to or 12 hours following the investigational product administration.
9. The subject received or is scheduled to receive a SPECT radiotracer within 24 hours prior to or 24 hours following the investigational product administration.
10. The subject received or is scheduled to receive a stress examination (other than the MR stress examination in this study) within 24 hours prior to or 24 hours following the investigational product administration.
11. The subject has experienced a myocardial infarction within the last 14 days.
12. The subject has experienced more than 1 previous myocardial infarction.
13. The subject has a bypass graft.
14. The subject has second or third degree atrioventricular block, sick sinus syndrome or a symptomatic bradycardia.
15. The subject suffers from asthma, bronchospasms or obstructive pulmonary disease.
16. The subject has severe hypotension (<90 mm Hg systolic).
17. The subject has unstable angina pectoris.
18. The subject has a decompensated congestive cardiac failure.
19. The subject's ECG shows a prolonged QT interval.
20. The subject has a contra-indication for MRI according to clinical guidelines, local regulations or manufacturer's recommendations.
21. The subject has cardiac arrhythmia considered by the investigator to be of a type or of a sufficient degree to make the subject unsuitable for the study.
22. The subject has consumed coffee, tea, coke, chocolate or other caffeinated beverages in the last 24 hours before the adenosine administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2003-07; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of perfusion CMR vs SPECT for sensitivity and specificity (binary reading) for the detection of coronary artery disease | SPECT and invasive angiography are performed within 4 weeks before or after CMR

SECONDARY OUTCOMES:
Assessment of the diagnostic performance of CMR and SPECT expressed as area under the receiver operator characteristics curve to detect coronary artery disease | SPECT and invasive angiography are performed within 4 weeks before or after CMR

CONTACTS AND LOCATIONS:
Overall Officials: Karoline Meurer, Med Vet, Study Director — Amersham Buchler GmbH & Co. KG, Ismaning b. Muenchen, Germany

REFERENCES:
- [Derived] Schwitter J, Wacker CM, Wilke N, Al-Saadi N, Sauer E, Huettle K, Schonberg SO, Debl K, Strohm O, Ahlstrom H, Dill T, Hoebel N, Simor T; MR-IMPACT investigators. Superior diagnostic performance of perfusion-cardiovascular magnetic resonance versus SPECT to detect coronary artery disease: The secondary endpoints of the multicenter multivendor MR-IMPACT II (Magnetic Resonance Imaging for Myocardial Perfusion Assessment in Coronary Artery Disease Trial). J Cardiovasc Magn Reson. 2012 Sep 2;14(1):61. doi: 10.1186/1532-429X-14-61. PMID 22938651